CLINICAL TRIAL: NCT05446350
Title: Modulating Speech Perception With Current Stimulation (SPEECHSTIM)
Brief Title: Modulating Speech Perception With Current Stimulation
Acronym: SPEECHSTIM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Toulouse (Other)
Collaborators: Centre National de la Recherche Scientifique, France (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: RC31/20/0340; 2020-A02707-32 (Other: Id-RCB); STIMPAROLE (Other: Acronyme)
Record Dates: First submitted 2022-07-01; First posted 2022-07-06 (Actual); Last update posted 2022-08-19 (Actual); Status verified 2022-08

CONDITIONS: Healthy
Keywords: Transcranial alternating current stimulation (tACS),; speech; perception; neural oscillations; entrainment; phase; neurofeedback
MeSH Terms: conditions — Speech | interventions — Transcranial Direct Current Stimulation; Neuroimaging

STUDY DESIGN:
Who Masked: Participant
Masking Description: masking to the conditions of the experiments
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Experiment 1 (Experimental): The aim of Experiment 1 is to understand how tACS operates on the neural level
  Interventions: Procedure: transcranial alternating current stimulation (tACS); Procedure: electroencephalography (EEG)
- Experiment 2 (Experimental): The aim of Experiment 2 is to increase efficacy of tACS and, consequently, its potential to play an important role in research and everyday life applications
  Interventions: Procedure: transcranial alternating current stimulation (tACS); Procedure: brain imaging (fMRI)
- Experiment 3 (Experimental): The aim of Experiment 3 is to reveal how tACS can boost speech perception in a multi-speaker scenario.
  Interventions: Procedure: transcranial alternating current stimulation (tACS)
- Experiment 4 (Experimental): The aim of Experiment 4 is to combine established techniques to create novel opportunities to improve speech perception
  Interventions: Procedure: transcranial alternating current stimulation (tACS); Procedure: electroencephalography (EEG) with neurofeedback

INTERVENTIONS:
Procedure: transcranial alternating current stimulation (tACS) — transcranial alternating current stimulation (tACS) used to manipulate how neural activity aligns to speech rhythm, leading to changes in speech perception
Procedure: electroencephalography (EEG) — analyse rhythmic electroencephalography responses that outlast the stimulation
  Arms: Experiment 1
Procedure: brain imaging (fMRI) — Using brain imaging (fMRI) to predict optimal stimulation protocols for individual participants
  Arms: Experiment 2
Procedure: electroencephalography (EEG) with neurofeedback — Using neurofeedback to teach participants to enhance their own neural entrainment
  Arms: Experiment 4

SUMMARY:
This study aims to further develop tACS as a tool to improve speech perception, by manipulation of brain-speech synchronisation ("entrainment"), thereby transforming a promising approach into a technique that can benefit to society on a large scale.

DETAILED DESCRIPTION:
Neural oscillations align their phase to the rhythm of speech. This phenomenon is termed neural entrainment and associated with successful speech comprehension. Importantly, we have demonstrated that transcranial alternating current stimulation (tACS) can be used to manipulate how neural activity aligns to speech rhythm, leading to changes in speech perception. The aim of Experiment 1 is to understand how tACS operates on the neural level. This aim will be reached by testing whether tACS produces rhythmic electroencephalography (EEG) responses that outlast the stimulation, indicating an involvement of endogenous oscillatory activity. The aim of Experiment 2 is to increase efficacy of tACS and, consequently, its potential to play an important role in research and everyday life applications. This aim will be reached by using brain imaging (fMRI) to predict optimal stimulation protocols for individual participants. The aim of Experiment 3 is to reveal how tACS can boost speech perception in a multi-speaker scenario. This aim will be reached by using tACS to enhance attended speech or suppress distracting speech, and by comparing these two approaches in their efficacy to boost speech perception. The aim of Experiment 4 is to combine established techniques to create novel opportunities to improve speech perception. This aim will be reached by using neurofeedback to teach participants to enhance their own neural entrainment, applying tACS to support them in this process.

ELIGIBILITY:
Inclusion Criteria:

* Subject aged between 18 and 50 years old
* informed written consent
* Absence of pro-epileptogenic drugs
* Absence of visual or hearing impairment incompatible with participation in the study

Exclusion Criteria:

* Pregnant or breastfeeding women,
* Persons protected by law adults under guardianship or curatorship
* Persons not affiliated to a Social Security scheme
* Subjects with progressive psychiatric or neurological pathology
* Subjects with a contraindication to tCS or MRI (history of epilepsy, severe head injury or brain/spinal cord surgery, cardiac pacemaker/defibrillator, implanted equipment activated by electrical, magnetic or mechanical system, hemostatic clip carriers of intracerebral aneurysms or carotid arteries, orthopedic implant carriers, claustrophobic, pregnancy).

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 126 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
correctly identified words | Day 1
  percentage of correctly identified words during or after tACS who will permit to evaluate efficacy of tACS to modulate speech perception and neural responses in different experimental conditions (involving electrophysiological, brain imaging, and perceptual measures)

SECONDARY OUTCOMES:
correctly identified words with different modality | day 1
  percentage of correctly identified words during or after tACS between different modality
oscillatory activities | Day 1
  measurement of oscillatory activities resulting from electrical stimulation: (frequency, power, and phase, latency) on the scalp and at the level of the sources and their synchronization with during or after tACS
neural activity | Day 1
  measurement of neural activity that results from electrical stimulation: fMRI (BOLD response) during or after tACS

CONTACTS AND LOCATIONS:
Overall Officials: Mathieu MARX, PU-PH, Principal Investigator — University Hospital, Toulouse
Locations (1):
- CHU Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] van Bree S, Sohoglu E, Davis MH, Zoefel B. Sustained neural rhythms reveal endogenous oscillations supporting speech perception. PLoS Biol. 2021 Feb 26;19(2):e3001142. doi: 10.1371/journal.pbio.3001142. eCollection 2021 Feb. PMID 33635855
- [Background] Zoefel B, Davis MH, Valente G, Riecke L. How to test for phasic modulation of neural and behavioural responses. Neuroimage. 2019 Nov 15;202:116175. doi: 10.1016/j.neuroimage.2019.116175. Epub 2019 Sep 6. PMID 31499178
- [Background] Zoefel B, Allard I, Anil M, Davis MH. Perception of Rhythmic Speech Is Modulated by Focal Bilateral Transcranial Alternating Current Stimulation. J Cogn Neurosci. 2020 Feb;32(2):226-240. doi: 10.1162/jocn_a_01490. Epub 2019 Oct 29. PMID 31659922